CLINICAL TRIAL: NCT05000463
Title: Ozone Therapy in Clinical, Psychological and Neurophysiological Pain Alleviation in Patients With Diabetic Neuropathy
Brief Title: Ozone Therapy in Patients With Diabetic Neuropathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB20025
Record Dates: First submitted 2021-08-04; First posted 2021-08-11 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2022-01

CONDITIONS: Pain, Chronic
MeSH Terms: conditions — Chronic Pain | interventions — Ozone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ozone group (Active Comparator): Ozone injection under ultrasound guidance in addition to the medical treatment
  Interventions: Drug: Ozone
- control group (Other): receive the medical treatment only. The medical treatment includes optimal glycemic control, vitamin B complex, a lipoic acid, selective serotonin reuptake inhibitors, and pregabalin
  Interventions: Drug: Convtrol group

INTERVENTIONS:
Drug: Ozone — The participants will lay flat and the area of injection will be prepared with antiseptic. Maintenance of ultrasonography probe sterility was also guaranteed using a sterile barrier. Under sonographic guidance, superficial peroneal nerve, deep peroneal, sural , asphenous, and tibila nerves will be injected An ozone/oxygen mixture ( 25μg/ml) will be injected in each nerev
  Arms: ozone group
Drug: Convtrol group — The medical treatment included optimal glycemic control, vitamin B complex, a lipoic acid, selective serotonin reuptake inhibitors, and pregabalin.
  Arms: control group

SUMMARY:
Diabetic neuropathies are the most prevalent chronic complications of diabetes mellitus. The early recognition and appropriate management of neuropathy in the patient with diabetes is important for patient's quality of life and life expectancy. Ozone is well known to have anti-inflammatory and analgesic effects through the inhibition of pro-inflammatory mediators; as well as. stimulation of anti-inflammatory mediators' release

DETAILED DESCRIPTION:
Introduction:

Diabetic neuropathies are the most prevalent chronic complications of diabetes mellitus. The early recognition and appropriate management of neuropathy in the patient with diabetes is important for patient's quality of life and life expectancy. The clinical symptoms of DPN range from pain and burning sensations (at rest or at night) to hypoesthesia, paresthesia, and/or numbness . Diabetic neuropathy can be axonal or demyelinating and can affect large or small neurons. Schwann cells, which are the most abundant glial cells, act as nerve axon insulators and modulators of neurobiology through their role in metabolic support and injury protection. In diabetic patients, church cells' function is disturbed, leading to loss of glial-axon communication and nerve homeostasis, which leads to fiber loss, neurodegeneration, and pain. Nerve conduction studies can detect these changes; however, there has been no effective therapy for the treatment of DPN until now.

Ozone is well known to have anti-inflammatory and analgesic effects through the inhibition of pro-inflammatory mediators; as well as. stimulation of anti-inflammatory mediators' release . Previous studies showed that Ozone promotes peripheral vascular integrity via induction of Vascular Endothelial Growth Factor (VEGF), Transforming Growth Factor Beta (TGF-β1) an Platelet-Derived Growth Factor (PDGF), according with the studies of Professor Bocci that demonstrated significantly increase and release of PDGF, TGF- β1 and VEGF in presence of Ozone .

ELIGIBILITY:
Inclusion Criteria:

* Sixty adult diabetic patients (type II DM)
* clinically symptomatized painful neuropathy for six or more months.

Exclusion Criteria:

* Patients with other causes of neuropathy (e.g., vitamin B12 deficiency), hereditary neuropathies and entrapment neuropathies, overt neuropathy with foot ulcers and/or amputation, peripheral vascular diseases, vertebral pathologies (e.g., previous surgery, foraminal stenosis, spinal canal stenosis, and/or vertebral disc herniation)
* Patients with other medical conditions such as connective tissue diseases, thyroid disorders, significant renal or hepatic dysfunction, platelet dysfunction syndrome, critical thrombocytopenia, hemodynamic instability and septicemia
* local infection at the site of the procedure
* Consistent use of nonsteroidal anti-inflammatory drugs within the last two weeks
* Systemic corticosteroid administration or local injection at the suspected treatment site within the last month
* Recent fever or illness, hemoglobin level <10 g/dL, platelet count <105 _ 109/L, and/or tobacco use.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-02-25 (Estimated); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-09-20 (Estimated)

PRIMARY OUTCOMES:
Pain Assessment | 6 months
  the visual analoge scale of pain (VAS) will be assessed. No pain VAS = 1, worst pain VAS= 10

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

REFERENCES:
- [Background] Bocci V, Zanardi I, Travagli V. Ozone: a new therapeutic agent in vascular diseases. Am J Cardiovasc Drugs. 2011;11(2):73-82. doi: 10.2165/11539890-000000000-00000. PMID 21446774
- [Background] Bril V, Tomioka S, Buchanan RA, Perkins BA; mTCNS Study Group. Reliability and validity of the modified Toronto Clinical Neuropathy Score in diabetic sensorimotor polyneuropathy. Diabet Med. 2009 Mar;26(3):240-6. doi: 10.1111/j.1464-5491.2009.02667.x. PMID 19317818
- [Background] Hassanien M, Elawamy A, Kamel EZ, Khalifa WA, Abolfadl GM, Roushdy ASI, El Zohne RA, Makarem YS. Perineural Platelet-Rich Plasma for Diabetic Neuropathic Pain, Could It Make a Difference? Pain Med. 2020 Apr 1;21(4):757-765. doi: 10.1093/pm/pnz140. PMID 31298289